CLINICAL TRIAL: NCT00254553
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Two Period Cross Over Trial to Validate Patient-Reported Outcome Measures for Use in Men With Late Onset Hypogonadism
Brief Title: A Study to Test a Measure of Symptoms of Older Men With Low Testosterone On and Off Testosterone Replacement Treatment (P05815)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment issues
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: P05815; P05815; 169001
Record Dates: First submitted 2005-11-14; First posted 2005-11-16 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Hypogonadism
MeSH Terms: conditions — Hypogonadism | interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator): Testim 1% (testosterone gel)
  Interventions: Drug: Testim 1% (testosterone gel)
- Arm 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Testim 1% (testosterone gel) — Testim_ 100 mg: two tubes of 50 mg of Testim_per day
  Other Names: Testim
  Arms: Arm 1
Drug: Placebo — two tubes of placebo per day
  Arms: Arm 2

SUMMARY:
Hypogonadal males, particularly those whose condition manifested later in life, may experience common symptoms associated with their hypogonadism. Questionnaires developed to assess these symptoms need to be tested. The primary purpose of this study is to test or validate the Patient-Reported Symptom Measure, Androgen Deficiency Quality of Life Questionnaire and the Patient Global Impression Scale.

ELIGIBILITY:
Inclusion Criteria:

Men with late-onset hypogonadism who are either on testosterone treatment or naïve of treatment:

* have symptoms of androgen deficiency at screening (after wash-out if applicable) i.e. with a positive score on the Androgen Deficiency in the Aging Male (ADAM) Questionnaire (a "yes" answer to questions 1 or 7 or any three other questions).
* morning total T levels of <=3 ng/mL (<=300 ng/dL; <=10.4 nmol/l) on two separate days prior to randomization (after appropriate wash-out, if applicable).
* calculated free T <=0.074 ng/mL.
* at least 50 and at most 75 years of age.
* BMI of at least 18 kg/m^2 or at most 32 kg/m^2

Inclusion Criteria for Normogonadal Men:

* morning total T levels <=3 ng/mL (<=300 ng/dL; <=10.4 nmol/L).
* calculated free T <=0.074 ng/mL.
* at least 50 and at most 75 years of age.
* BMI of at least 18 kg/m^2 or at most 32 kg/m^2

Exclusion Criteria:

* History or current diagnosis of prostate cancer or any clinically significant finding on prostate examination
* Severe obstructive symptoms of benign prostate hypertrophy
* Prostate specific antigen (PSA) levels greater than 4 ng/mL at screening
* History or current diagnosis of carcinoma of the breast
* Known chronic polycythemia and/or hematocrit greater than 50% at screening
* Treatment-naïve subjects with hyperprolactinemia at screening (serum prolactin level >=50 ng/mL)
* Hematological or biochemical values at screening outside the reference ranges considered as clinically significant in the opinion of the investigator
* clinically significant abnormal physical finding prior to randomization
* sensitive to trial medication or its components
* History or presence of hepatic or renal disorder considered as clinically relevant in the opinion of the investigator.

Exclusion Criteria for Normogonadal Men:

* Presence or previous diagnosis of androgen deficiency.
* Previous or present use of testosterone preparations
* Use of medication within the 12 weeks prior to the visit that may interfere with the objectives of the trial: hypothalamic/pituitary hormones and analogues (e.g., gonadotropins, ACTH, STH, Gn-RH agonists and antagonists, etc.); sex steroid
* Any other disease that in the opinion of the investigator might compromise or confound the subject's symptomatology (e.g., presence of clinically significant depression or other psychiatric disorders, unstable endocrine disorder, sleep apnea, cardiovascular and cerebrovascular diseases, etc.)

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2005-07; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Patient -reported outcome measures | Baseline and after six weeks of treatment or placebo